CLINICAL TRIAL: NCT01087164
Title: Brief Interventions to Increase HPV Vaccine Acceptance in School-based Health Centers in Adolescents
Brief Title: Brief Interventions to Increase HPV Vaccine Acceptance in School-based Health Centers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indiana University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Vaughn Rickert, Professor and Director, Section of Adolescent Medicine, Indiana University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0911-50
Record Dates: First submitted 2009-02-02; First posted 2010-03-16 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Human Papillomavirus Infection
Keywords: Vaccine acceptance; human papillomavirus; brief messages; social compliance; Message sidedness
MeSH Terms: conditions — Papillomavirus Infections | interventions — Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compliance (Experimental): Parents will be randomized to receive high or no compliance condition where those in the experimental group will be asked about whether or not they will protect their daughter from cervical cancer or for males, their son from genital warts.
  Interventions: Behavioral: Compliance
- Message sidedness (Experimental): Parents will be given either a one-sided verbal message or a two-sided verbal message about the HPV vaccine.
  Interventions: Behavioral: Message sidedness

INTERVENTIONS:
Behavioral: Compliance — Parent will either receive a high or no compliance condition where each is asked to endorse the importance of prevention cervical cancer or genital warts depending on their teen's gender.
  Arms: Compliance
Behavioral: Message sidedness — Parent will receive either a one-sided or two-sided message about the HPV vaccine
  Arms: Message sidedness

SUMMARY:
Using health behavior theories and theories related to the effects of persuasive messages (i.e., inoculation theory), we plan to: 1. Systematically test the effects of brief persuasive message interventions on receipt of the first dose of HPV vaccine; and 2. evaluate the effects of the interventions on followup with subsequent doses of vaccine (using reminder notices with persuasive message content). One set of interventions will involve a comparison of a 1 sided message, which only emphasizes the positive aspects of a recommended behavior, with a 2 sided message, which presents negative aspects of the behavior followed by positive counterarguments. A second set of interventions will involve a test of a social compliance (foot-in-the-door technique, in which half of the parent participants will be asked to respond to a high compliance request (i.e., a request likely to generate high compliance, such as, "Do you want to protect your daughter from cancer? or for male children, "Do you want to protect your son from genital warts?"before subsequently being asked about actually having their adolescents vaccinated. The other half of the parents will not receive a high compliance request. Parents of 11-14 year old adolescents will be randomized to the two sets of interventions, resulting in a 2 X 2 design: message sidedness (1 sided; 2 sided) and social compliance request (yes; no). The specific aims of this proposal are to evaluate the 1) efficacy of 2 sided vs. 1 sided messages on rates of HPV vaccination; 2) the efficacy of a social compliance intervention on rates of HPV vaccination; and 3) potential moderators and mediators of message effect on vaccine acceptance.

DETAILED DESCRIPTION:
The proposed study will employ a randomized, full factorial experimental design to examine the effects of brief message interventions on parents' acceptance of the first dose of HPV vaccine for their adolescents aged 11-14 years, as well as follow through with subsequent doses. Specifically, the study will employ a 2 x 2 experimental design, in which participants will be assigned randomly to one of two different message sidedness conditions (1 sided vs. 2 sided) and two social compliance conditions (high compliance request [HCR] vs. noHCR). The interventions will be administered by a bilingual research assistant who will read, verbatim, scripts provided to them. Computer assisted telephone interview (CATI) will be used to gather demographic and background information as well as parental health beliefs regarding preexisting worries about HPV vaccine leading to safety concerns (moderator variable) prior to administration of the interventions. After the interventions, additional health beliefs will be assessed (mediators).

1. A greater proportion of girls as compared to boys will receive a first dose of vaccine.
2. Among both girls and boys who receive a first dose of Gardasil™, no differences in completion rates will be detected.
3. The social compliance intervention to be more effective with parents of girls as compared to parents of boys. This prediction of a differential effect is based on the fact that cervical cancer will be seen as a more serious and less stigmatizing condition than genital warts.

In summary, the implementation of this protocol will allow us to systematically examine the use of two different interventions on parents of both boys and girls. Thus, parents (n=800) of 11-14 year old girls and boys will be randomized to the two sets of interventions, resulting in a 2 X 2 design: message sidedness (1-sided; 2-sided) and HCR (yes; no).

ELIGIBILITY:
Inclusion Criteria:

* The parents of adolescent males and females (aged 11-14 years) who have provided written consent for their adolescent to receive health care services through the Teen Health Center, Inc, a nonprofit organization that works in collaboration with the Department of Pediatrics at the University of Texas Medical Branch, Galveston, Texas and whose adolescents have not received their first dose of HPV vaccine, will be eligible to participate.

Exclusion Criteria:

* Having received one or more doses of the HPV vaccine Gardasil

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Gardasil immunization | One year
  Parent signs vaccine information sheet and returns to school-based health center. Adolescent is vaccinated with first dose of Gardasil by licensed health care professional.

SECONDARY OUTCOMES:
Completion of three dose series of Gardasil | Three years
  We will identify all enrolled parents to determine whether their adolescent received all three required Gardasil immunization across a three year period.
Message type | Two years
  Determine whether the type of message delivered to parent, i.e., one-sided or two-sided, increases the number of first dose immunizations.
Gender | One year
  Determine if there are gender differences between male and female children relative to first dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Vaughn I Rickert, PsyD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Teen Health Centers, Galveston, Texas, United States

REFERENCES:
- [Result] Rickert VI, Auslander BA, Cox DS, Rosenthal SL, Rickert JA, Rupp R, Zimet GD. School-based vaccination of young US males: impact of health beliefs on intent and first dose acceptance. Vaccine. 2014 Apr 7;32(17):1982-7. doi: 10.1016/j.vaccine.2014.01.049. Epub 2014 Jan 31. PMID 24492015